CLINICAL TRIAL: NCT06217055
Title: Comparison of Remimazolam-based Monitored Anesthesia Care With Inhalation General Anesthesia Under the Guidance of an ANI Monitor During TURB: a Randomized Controlled Trial
Brief Title: Comparison of Remimazolam-based MAC With Inhalation General Anesthesia Under the Guidance of an ANI Monitor During TURB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-1206
Record Dates: First submitted 2023-11-22; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Patients Undergoing Transurethral Resection of Bladder
MeSH Terms: interventions — Anesthesia, General; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remimazolam based MAC group (Experimental): remimazolam based monitored anesthesia care
  Interventions: Drug: remimazolam based MAC
- inhalation general anesthesia group (Active Comparator): general anesthesia with sevoflurane
  Interventions: Drug: general anesthesia with sevoflurane

INTERVENTIONS:
Drug: remimazolam based MAC — The surgery will be performed under monitored anesthesia care by maintaining spontaneous breathing using remimazolam.
  Arms: remimazolam based MAC group
Drug: general anesthesia with sevoflurane — The surgery will be performed under mechanical ventilation with inhalation general anesthesia
  Arms: inhalation general anesthesia group

SUMMARY:
In patients undergoing transurethral resection of bladder, the effect of remimazolam-based monitored anesthesia care (MAC) and inhalational general anesthesia will be compared under guidance by analgesia nociception index (ANI) monitoring. Anesthesia time, operation time, anesthesia time excluding operation time and total dose of opioid will be compared.

DETAILED DESCRIPTION:
In remimazolam-based MAC group, anesthesia will be induced with remimazolam and spontaneous breathing will be maintained. The dose of remimazolam and remifentanil will be adjusted according to the patient state index (PSI) and the analgesia nociception index(ANI).

In inhalation general anesthesia group, anesthesia will be induced with propofol and rocuronium and maintained with sevoflurane and remifentanil. Mechanical ventilation will be maintained by inserting laryngeal mask airway (LMA) or endotracheal tube. The doses of sevoflurane and remifentanil will be adjusted according to the patient state index (PSI) and the analgesia nociception index(ANI).

Surgery cost, anesthesia cost, patient and surgeon's satisfaction score, pain score, PONV score and the incidence of hypotension and hypoxemia will be compared.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing transurethral bladder resection

Exclusion Criteria:

* ASA class 4
* emergency surgery
* history of hypersensitivity to sevoflurane, propofol and remimazolam
* galactose intolerance
* patient refusal
* patients in whom muscular relaxation are needed.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
anesthesia time excluding operation time | 0-1 hour after the end of surgery (Time point at which patient exit the operating room)
  anesthesia time excluding operation time

SECONDARY OUTCOMES:
surgery cost and anesthesia cost | 1 month after surgery
  surgery cost and anesthesia cost: insured cost and non-insured cost
surgeon's satisfaction score | At the end of surgery
  surgeon's satisfaction score: very poor (1)/ poor (2)/ satisfactory (3)/ good (4)/excellent (5)
patient's satisfaction score | 0-2 hour after surgery (Time points at patient discharge from recovery room)
  patient's satisfaction score: very poor (1)/ poor (2)/ satisfactory (3)/ good (4)/excellent (5)
pain score | 0-2 hour after surgery (Time points at patient discharge from recovery room), and 6 hour after surgery
  pain score : NRS 0-10 The numerical rating scale requires the patient to rate their pain or nausea/vomiting on a defined scale. Numerical rating scale (NRS) is the simplest and most commonly used scale. The numerical scale is most commonly 0 to 10, with 0 being "no pain or no nausea/vomiting" and 10 being "the worst pain or nausea/vomiting imaginable.
PONV score | 0-2 hour after surgery (Time points at patient discharge from recovery room), and 6 hour after surgery
  PONV was defined as nausea or vomiting score.
incidence of hypotension | At the end of surgery
  hypotension: baseline BP reduction (20%)
incidence of hypoxemia | At the end of surgery
  hypoxemia : unresponsive to a jaw thrust maneuver and SPO2 <92%

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university college of medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided